CLINICAL TRIAL: NCT06831539
Title: Impact of PEG Bowel Preparation on Gut Microbiome Composition Recovery
Acronym: PEG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-12213
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Healthy Participants
Keywords: PegLyte; Microbiome
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm study evaluating the impact of PEG bowel preparation on the gut microbiome in volunteer participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer participant cohort (Experimental): For healthy volunteer participants, PEG bowel preparation will be administered and participants will collect stool samples before and after PEG at specified timepoints.
  Interventions: Drug: PEGLyte bowel preparation

INTERVENTIONS:
Drug: PEGLyte bowel preparation — Volunteers will be administered 4L of PEG bowel preparation. The following instructions will be provided with the prescription:
  1. Fill the supplied container containing the bowel cleanse powder with lukewarm water (to facilitate dissolution) to the 4-liter fill line. The solution is clear and colourless when reconstituted to a final volume of 4 liters.
  2. After capping the container, shake vigorously several times to ensure that the ingredients are dissolved. The solution is more palatable if chilled prior to drinking. When reconstituted use within 48 hours.
  3. Attempt to drink a maximum of 4 liters at a rate of 240 mL (8 oz.) every 10 minutes, until 4 liters has been consumed or the rectal effluent is clear. Rapid drinking of each portion is preferred to drinking small amounts continuously.
  4. The first bowel movements should occur approximately one hour after the start of bowel cleanse administration. Continue drinking until the watery stool is clear and free of solid matter.
  Other Names: PEG

SUMMARY:
The main objective is to evaluate the impact of intestinal preparation on the composition, diversity and metabolome of the intestinal microbiota.

DETAILED DESCRIPTION:
Based on the limited literature that PEG does not significantly impact the microbiome, certain investigators ascertain that administration of PEG without any subsequent FMT would represents the gold-standard control group. On the other hand, other investigators raised their concern that perturbation of the microbiome with PEG without subsequent replacement with FMT might negatively impact immune checkpoint inhibitor efficacy. Therefore, there is an unmet need to conduct a study using the metagenomic shotgun sequencing to precisely understand the impact of bowel preparation on gut microbiome composition and on the dynamics of recovery of the gut microbiome after bowel preparation to better design microbiome-centered trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer participant cohort:

  1. > 18 years of age
  2. The participant has provided documented informed consent for the participation and to complete PEG bowel preparation and return collected stool samples.

Exclusion Criteria:

* An ileus
* Significant gastric retention
* Suspected or established mechanical bowel obstruction
* Inflammatory or infectious gastrointestinal condition
* Neurologic or cognitive impairment that prevents safe swallowing
* Recent history (<1 year) of cancer that still requires ongoing treatment
* Recent use of antibiotics 1 month prior to participation in the trial
* History of cardiac disease
* History of active renal dysfunction
* Presence of any absolute contraindication to PEG bowel preparation according to manufacturer labeling

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of bowel preparation on the gut microbiota at 1 week after bowel preparation. | At week 1
  Study of the gut microbiota composition at 1 week after bowel preparation.

SECONDARY OUTCOMES:
Gut microbiome composition, diversity, and gut metabolome profile at 1 month and 3 months after bowel preparation | At 1 month and 3 months
  1. Gut metabolite composition at 1 month after bowel preparation.
  2. Gut microbiota composition, diversity, metabolite composition at 1 month and 3 months after bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Elkrief, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada